CLINICAL TRIAL: NCT06044779
Title: Transversus Abdominis Plane (TAP) Block and Erector Spinae Plane (ESP) Block Comparison on Postoperative Pain and the Need for Morphine in Gynecological Surgery Patients Who Underwent Median Incision in Hasan Sadikin General Hospital
Brief Title: TAP vs. ESP Block for Gynecological Post Operative Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universitas Padjadjaran (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: AN-202309.03
Record Dates: First submitted 2023-09-10; First posted 2023-09-21 (Actual); Last update posted 2023-09-22 (Actual); Status verified 2023-09

CONDITIONS: Nerve Block; Pain, Postoperative
Keywords: Transversus Abdominis Plane Block; Erector Spinae Plane Block; Postoperative Pain; Gynecological Surgery
MeSH Terms: conditions — Pain, Postoperative | interventions — Bupivacaine

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Transversus Abdominis Plane (TAP) Anesthestic Block (Active Comparator): Ultrasound-guided TAP block is done using 20 mL of 0.25% Bupivacaine administered at the lateral abdominal wall between the costal margin and the iliac crest
  Interventions: Procedure: Transversus Abdominis Plane Block using 0.25% Bupivacaine
- Erector Spinae Plane (ESP) Anesthetic Block (Active Comparator): Ultrasound-guided ESP block is done using 20 mL of 0.25% Bupivacaine administered at the tip of the transverse process at the T9 level
  Interventions: Procedure: Erector Spinae Plane Block using 0.25% Bupivacaine

INTERVENTIONS:
Procedure: Transversus Abdominis Plane Block using 0.25% Bupivacaine — TAP block regional anesthesia with ultrasound guidance with administration of 20 mL of 0.25% Bupivacaine in the abdominal wall before the operation is completed. The patient was also fitted with a morphine PCA device with a background dose of 5 µg/kgBW/hour and a rescue dose of 1 mg with a lockout interval of 10 minutes.
  Arms: Transversus Abdominis Plane (TAP) Anesthestic Block
Procedure: Erector Spinae Plane Block using 0.25% Bupivacaine — Regional anesthesia ESP block under ultrasound guidance with 20 mL of 0.25% bupivacaine at the tip of the transverse process at the T9 level before completion of surgery. The patient was also fitted with a morphine PCA device with a background dose of 5 µg/kgBW/hour and a rescue dose of 1 mg with a lockout interval of 10 minutes.
  Arms: Erector Spinae Plane (ESP) Anesthetic Block

SUMMARY:
The goal of this double blind randomized controlled trial is to compare transversus abdominis plane block and erector spinae plane block in gynecological surgery patients. The main questions it aims to answer are:

* What are the numerical post-operative pain scores in these two groups?
* Is there any significant difference in the numerical post-operative pain scores between subjects who underwent TAP block and subjects who underwent ESP block?
* What are the differences in the time needed for additional morphine in these two groups?
* Is there any significant differences in the time needed for additional morphine between subjects who underwent TAP block and subjects who underwent ESP block?

ELIGIBILITY:
Inclusion Criteria:

* Subjects with gynecological surgery techniques with a median incision include: hysterectomy, myomectomy, salpingectomy, ovarectomy and ovarian cystectomy.
* Subjects with physical status based on the American Society of Anesthesiologists (ASA) in categories I-II
* Subjects who are willing to sign informed consent form.

Exclusion Criteria:

* The patient has a history of allergies to local anesthetic drugs used for TAP blockade or ESP blockade and is allergic to morphine.
* Patients who have skin infections at the injection site.
* Patients with a history of chronic pain, namely a history of pain for more than 1 month obtained from history taking.
* Patients with a history of chronic pain treatment obtained from history taking.
* Patients with impaired kidney function (Ureum >39 mg/dL; Creatinine >1.3 mg/dL) and liver (SGOT >37 U/L; SGPT >59 U/L), myopathy, coagulopathy obtained from the results of supporting examinations, heart rhythm disorders obtained from the results of an EKG examination and neurological disorders in the form of hypesthesia or paraesthesia obtained from the results of a physical examination in the form of a sensory examination.
* The patient is pregnant as determined by history taking.
* Patients who are illiterate as obtained from history taking.
* The patient was uncooperative during examination.

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Female
Enrollment: 40 (Actual)
Dates: Start 2022-12-27 (Actual); Primary Completion 2023-03-26 (Actual); Study Completion 2023-03-26 (Actual)

PRIMARY OUTCOMES:
Postoperative Numerical Rating Scale | 24 hours post operative
  The degree of pain assessment is classified based on the Numeric Rating Scale pain assessment scale) with the lowest scale being no pain (value 0), up to the heaviest pain scale (value 10) when still, namely when the patient does not make any movement and moves, namely when mobilization is carried out on the left side and right tilt

SECONDARY OUTCOMES:
Total postoperative morphine requirements | 24 hours post operative
  The total amount of morphine required by study subjects over 24 hours to reduce postoperative pain
Time of first need for analgesic rescue | 24 hours post operative
  The time required by study subjects to press the PCA to obtain analgesics was first calculated from the time it was installed in the recovery room

CONTACTS AND LOCATIONS:
Overall Officials: Doddy M Tavianto, MD, Study Director — Faculty of Medicine Universitas Padjadjaran Bandung; Osmond M Pison, MD, Study Director — Faculty of Medicine Universitas Padjadjaran Bandung; Azka P Rakhimulllah, MD, Principal Investigator — Faculty of Medicine Universitas Padjadjaran Bandung
Locations (1):
- Hasan Sadikin General Hospital, Bandung, West Java, Indonesia